CLINICAL TRIAL: NCT01906411
Title: Dopaminergic Function and Food Reward
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Dr., University Hospital Tuebingen
Other Study IDs: DAD
Record Dates: First submitted 2013-07-08; First posted 2013-07-24 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Adiposity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subjecst with different BMI
  Interventions: Dietary Supplement: Dopamine depletion vs. Balanced aminoacid drink

INTERVENTIONS:
Dietary Supplement: Dopamine depletion vs. Balanced aminoacid drink

SUMMARY:
The broad aim of the study is to obtain a better understanding of alterations in mesolimbic reward pathways in adiposity based on the hypothesis of a hypofunctioning reward system in obesity.

This will be achieved by integrating a functional neuroimaging (fMRI) with behavioral reward tasks and the modulation of the dopamine level by dopamine depletion.

ELIGIBILITY:
Inclusion Criteria:

* female
* healthy

Exclusion Criteria:

* fMRI contraindications
* claustrophobia

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Differential brain functions in the dopaminergic reward system | 4 hours after intake of the dopamine depletion or balanced aminoacid drink
  differential brain fuctions will be measured by blood oxygen level dependent effect.

SECONDARY OUTCOMES:
amino acid level changes due to dopamine depletion | 4 hours after intake of the dopamine depletion or balanced aminoacid drink

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, MEG Center, Tübingen, Germany